CLINICAL TRIAL: NCT01911312
Title: Evaluation of Thermal-Aided Muscle Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Niveus Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLP3.00
Record Dates: First submitted 2013-07-12; First posted 2013-07-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Weakness; Atrophy
MeSH Terms: conditions — Asthenia; Atrophy

ARMS (2):
- Intervention (Experimental)
  Interventions: Device: Thermal-aided muscle stimulation
- Body Temperature Control (Active Comparator): Stimulation performed with body temperature control
  Interventions: Device: Body Temperature Stimulation

INTERVENTIONS:
Device: Thermal-aided muscle stimulation — Thermal-aided muscle stimulation is applied to subject quadriceps (one leg) with Niveus Medical Muscle Stimulation System 110
  Arms: Intervention
Device: Body Temperature Stimulation — Body temperature stimulation is applied to subject quadriceps (one leg) with Niveus Medical Muscle Stimulation System 110
  Arms: Body Temperature Control

SUMMARY:
An investigation into the relative effectiveness of thermal-aided muscle stimulation vs. body temperature muscle stimulation for eliciting muscle contraction in the quadriceps

ELIGIBILITY:
Inclusion Criteria:

* Subject does not meet any exclusion criteria

Exclusion Criteria:

* Age < 18 years
* Subject is pregnant
* Subject has an implanted pacemaker/defibrillator
* Subject diagnosed with epilepsy
* Subject has implanted metallic femoral rods
* Subject is chair- or bed-bound
* Subject has neuromuscular disease or abnormalities
* Subject BMI > 45
* Evidence of disease or condition that, in the opinion of the investigator, may compromise the conduct of or results of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-07; Primary Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Muscle Contraction Force | At 30 s intervals for 20 minutes
  Measured in Newtons

CONTACTS AND LOCATIONS:
Locations (1):
- Melchor Pavilion, Mountain View, California, United States